CLINICAL TRIAL: NCT07356648
Title: Investigation of the Effectiveness of Diadynamic Current in Patients With Carpal Tunnel Syndrome
Brief Title: Diadynamic Current and Carpal Tunnel Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Decision No: 2025/69
Record Dates: First submitted 2025-12-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Diadynamic Current; Electrotherapy; Pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Diadynamic Current Plus Splint (Experimental): Diadynamic current (DDC) is a routine physical therapy modality applied in the physical medicine and rehabilitation clinic to reduce symptoms in various conditions. In individuals with carpal tunnel syndrome (CTS), splinting is routinely prescribed as a first-line conservative treatment. In addition, physical therapy modalities such as DDC are applied in cases where adequate benefit is not achieved with splint therapy alone.
  Since splinting is provided as the initial conservative treatment in routine clinical practice, no delay or loss of treatment time occurs. Individuals receiving splint therapy are informed about DDC treatment, and those providing consent for 10 physical therapy sessions are allocated to the DDC group.
  Interventions: Procedure: Diadynamic Current
- Group 2: Splint-Only Group (Active Comparator): In individuals with carpal tunnel syndrome, splinting is routinely prescribed as a first-line conservative treatment.
  Interventions: Procedure: Diadynamic Current; Procedure: Wrist Splint

INTERVENTIONS:
Procedure: Diadynamic Current — Diadynamic current (DDC) is a routine therapeutic modality applied in the physical medicine and rehabilitation clinic to alleviate symptoms in various conditions. In individuals with carpal tunnel syndrome (CTS), DDC is routinely administered in cases where sufficient benefit is not achieved with splinting and transcutaneous electrical nerve stimulation (TENS).
  For this purpose, diadynamic current is applied to the palmar surface of the hand and the volar surface of the forearm using equal-sized carbon electrodes (6 × 6 cm). A sequence of different types of diadynamic currents is administered for a total duration of 10 minutes as follows: diphase fixe (DF) for 2 minutes, monophase fixe (MF) for 3 minutes, longues périodes (LP) for 3 minutes, and courtes périodes (CP) for 2 minutes.
  The treatment duration, parameters, and sequence of diadynamic currents are based on Bernard's current methodology and are identical to the procedure described by Ratajczak et al.
Procedure: Wrist Splint — In individuals with carpal tunnel syndrome, splinting is routinely prescribed as a first-line conservative treatment. A resting wrist splint extending from the distal forearm to the hand and maintaining the wrist in a neutral position is provided to both groups. The splint is worn every night before bedtime, maintained throughout the night, and removed in the morning upon waking.
  Arms: Group 2: Splint-Only Group

SUMMARY:
Carpal tunnel syndrome (CTS), first described by Paget in 1854, is the most common entrapment neuropathy. Conservative treatment approaches are prioritized in patients with mild to moderate CTS. Conservative management includes education, tendon and median nerve gliding exercises, physical therapy modalities, kinesiotaping, manual therapy techniques, injection options, and oral medical treatments. First-line treatment generally consists of education, exercise, and splinting.

Tendon and median nerve gliding exercises represent key components of conservative treatment. Splinting is recommended at all stages of CTS, with wrist splints designed to maintain a neutral position being the most commonly preferred option. The prevailing approach in the literature supports the use of splints primarily during nighttime.

Diadynamic current (DDC) is considered to have a composite analgesic mechanism, primarily explained by the gate control theory. Additional mechanisms suggest that DDC affects both sensory and motor nerves and may increase endorphin release, contributing to pain relief. A single treatment session typically does not exceed 12 minutes. Some studies indicate that the analgesic effect of DDC may be greater than that of transcutaneous electrical nerve stimulation (TENS). Although TENS is widely used in physical therapy and rehabilitation practice, DDC may represent a realistic alternative for clinical pain management.

The aim of the study is to evaluate the effect of diadynamic current therapy on clinical symptoms in patients with CTS and to investigate its impact on electrophysiological findings of the median nerve.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and electrophysiologically diagnosed with carpal tunnel syndrome (CTS)
* Provision of informed consent
* Age between 18 and 65 years

Exclusion Criteria:

* Age below 18 years or above 65 years
* Median nerve distal motor latency > 6.0 ms on nerve conduction studies (NCS)
* Thenar muscle atrophy
* History of carpal tunnel syndrome surgery
* History of steroid injection into the carpal tunnel
* History of physical therapy for CTS within the past 6 months
* Cervical radiculopathy
* Tenosynovitis in the ipsilateral upper extremity
* Other compressive neuropathy in the ipsilateral upper extremity
* Peripheral polyneuropathy
* History of trauma or fracture involving the hand, wrist, or forearm
* Pregnancy
* Presence of metabolic disease
* Inflammatory rheumatic disease
* Acute and/or chronic renal failure
* Severe cognitive impairment preventing understanding and following simple instructions
* Severe visual or hearing impairment preventing participation in treatment
* Current use of pregabalin or gabapentin
* Systemic diseases (e.g., diabetes mellitus, hypothyroidism, rheumatic diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Boston Carpal Tunnel Questionnaire Symptom Severity Scale Score | Baseline and 6 weeks
  Boston Carpal Tunnel Questionnaire - Symptom Severity Scale (BCTQ-SSS) is a patient-reported outcome measure assessing symptom severity in individuals with carpal tunnel syndrome. Scores range from 1 to 5, with higher scores indicating worse symptom severity.
Change from Baseline in Boston Carpal Tunnel Questionnaire Functional Status Scale Score | Baseline and 6 weeks
  Boston Carpal Tunnel Questionnaire - Functional Status Scale (BCTQ-FSS) assesses functional status and difficulty in daily activities in individuals with carpal tunnel syndrome. Scores range from 1 to 5, with higher scores indicating worse functional status.
Change from Baseline in Hand Grip Strength (kg) | Baseline and 6 weeks
  Hand Grip Strength was measured using a Saehan SH5001 Hydraulic Hand Dynamometer and recorded in kg. Higher values indicate greater grip strength.
Change from Baseline in Pinch Grip Strength (kg) | Baseline and 6 weeks
  Pinch Grip Strength was measured using a Saehan SH5005-1 Mechanical Pinch Gauge and recorded in kg. Higher values indicate greater pinch strength.
Electrophysiological Assessment-Median Distal Motor Latency | Baseline and 6 weeks
  Median distal motor latency was evaluated using nerve conduction studies (NCS) performed at the Electromyography Laboratory of the Department of Neurology, Düzce University Faculty of Medicine. Measurements were recorded in milliseconds (ms).
  Electrophysiological carpal tunnel syndrome was defined as median distal motor latency ≥ 4.0 ms.
Electrophysiological Assessment- Median Sensory Nerve Conduction Velocity | Baseline and 6 weeks
  Median sensory nerve conduction velocity was evaluated using nerve conduction studies (NCS) performed at the Electromyography Laboratory of the Department of Neurology, Düzce University Faculty of Medicine. Measurements were recorded in meters per second (m/s).
  Electrophysiological carpal tunnel syndrome was defined as median sensory nerve conduction velocity ≤ 40 m/s.
Electrophysiological Assessment-Median-Ulnar Sensory Peak Latency Difference | Baseline and 6 weeks
  Comparative median-ulnar sensory peak latency analysis was performed using fourth-digit recordings with wrist stimulation during nerve conduction studies (NCS). Measurements were recorded in milliseconds (ms).
  Electrophysiological carpal tunnel syndrome was defined as median sensory peak latency from the fourth digit exceeding ulnar latency by ≥ 0.4 ms.

CONTACTS AND LOCATIONS:
Locations (1):
- Düzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Demidas A, Zarzycki M. Touch and Pain Sensations in Diadynamic Current (DD) and Transcutaneous Electrical Nerve Stimulation (TENS): A Randomized Study. Biomed Res Int. 2019 Jul 17;2019:9073073. doi: 10.1155/2019/9073073. eCollection 2019. PMID 31380442
- [Result] Koca I, Boyaci A, Tutoglu A, Ucar M, Kocaturk O. Assessment of the effectiveness of interferential current therapy and TENS in the management of carpal tunnel syndrome: a randomized controlled study. Rheumatol Int. 2014 Dec;34(12):1639-45. doi: 10.1007/s00296-014-3005-3. Epub 2014 Apr 12. PMID 24728028

DOCUMENTS (1):
  • Study Protocol (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT07356648/Prot_000.pdf